CLINICAL TRIAL: NCT00939991
Title: Phase I/II Study of Bevacizumab Plus Daily Temozolomide and Vorinostat for Recurrent Malignant Glioma Patients
Brief Title: Suberoylanilide Hydroxamic Acid (SAHA), Bevacizumab, Daily Temozolomide for Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Katy Peters (Other)
Collaborators: Genentech, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Katy Peters, Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00016446
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-05

CONDITIONS: Brain Tumor; Glioblastoma
Keywords: GBM
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma | interventions — Bevacizumab; Temozolomide; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Phase I- Bevacizumab will be administered intravenously every other week. Temozolomide will be administered on a continuous daily dosing schedule. Vorinostat will be administered daily on days 1-7 and 15-21 of each 28 day cycle. The dose of Vorinostat will be escalated in successive cohorts of patients to determine the MTD of this regimen.
  Interventions: Drug: Vorinostst/Bevacizumab/Temozolomide

INTERVENTIONS:
Drug: Vorinostst/Bevacizumab/Temozolomide — Bevacizumab will be administered intravenously at the dose 10 mg/kg every other week. Temozolomide will be administered on a continuous daily dosing schedule at 50 mg/m2/day. Vorinostat will be administered daily on days 1-7 and 15-21 of each 28 day cycle. The dose of Vorinostat will be escalated in successive cohorts of patients to determine the MTD of this regimen. Bevacizumab doses may be given by the local oncologists under the direction of the Duke investigators.
  Other Names: Bevacizumab (Avastin); Temozolomide (Temodar); Vorinostat (Zolinza)

SUMMARY:
This is a Phase I/II open-label, single-arm study among recurrent malignant glioma patients. Patients will be treated with Vorinostat in combination with Bevacizumab (BV) (10 mg/kg) and Temozolomide (T) (50 mg/m2/day) BV is administered every 2 weeks. Temozolomide will be taken orally once every day. Vorinostat will be taken orally on days 1-7 and 15-21 of each 28-day cycle. In the phase I portion of this study, the dose of Vorinostat will be escalated in successive cohorts of patients to determine the maximum tolerated dose (MTD) based on dose-limiting toxicities (DLTs). In the phase II portion of this study, the dose of Vorinostat will be the MTD determined in the phase I portion. The primary endpoint of the phase II study is 6-month progression-free survival (PFS) for recurrent GBM (Glioblastoma) patients. This study will be conducted at The Preston Robert Tisch Brain Tumor Center at Duke.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of malignant glioma and radiographic evidence of recurrence or disease progression (defined as either a greater than 25% increase in the largest bidimensional product of enhancement or a new enhancing lesion) following prior therapy. In addition, the following must be met:

Phase I specific

* WHO grade 3 or 4 malignant glioma Phase II specific
* WHO grade 4 malignant glioma
* No more than 2 prior episodes of disease progression

Common to both Phase I and Phase II

* Age * 18 years
* KPS (Karnofsky Performance Scale) ≥ 70%
* An interval of at least 4 weeks between prior surgical resection or one week from stereotactic biopsy
* An interval of at least 12 weeks from the end of prior radiotherapy unless there is a new area of enhancement consistent with recurrent tumor outside of the radiation field, or there are progressive changes on MRI on at least two consecutive MRI scans at least four weeks apart, or there is biopsy-proven tumor progression
* An interval of at least 4 weeks from prior chemotherapy (6 weeks for nitrosoureas) or investigational agent unless the patient has recovered from all anticipated toxicities associated with that therapy
* Hematocrit ≥ 29%, ANC ≥ 1,000 cells/*l, platelets ≥ 100,000 cells/*l
* Serum creatinine < 1.5 times upper limit of normal, serum SGOT < 2.5 times upper limit of normal and bilirubin < 2.0 times upper limit of normal
* Signed informed consent approved by the Institutional Review Board prior to patient entry
* No evidence of hemorrhage on the baseline MRI or CT scan other than those that are stable grade 1
* If sexually active, patients will take contraceptive measures for the duration of the treatments. Medically acceptable contraceptives include:

  1. surgical sterilization (such as a tubal ligation, hysterectomy, vasectomy),
  2. approved hormonal contraceptives (such as birth control pills, patches, implants or injections),
  3. barrier methods (such as a condom or diaphragm) used with a spermicide, or
  4. an intrauterine device (IUD).

Exclusion Criteria:

* Prior therapy with histone deacetylase inhibitors; valproic acid is not permitted and patients previously treated with valproic acid must be off valproic acid for at least 30 days prior to initiation of study medication
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids
* Active infection requiring intravenous antibiotics
* Progression on prior bevacizumab or daily temozolomide
* Grade 3 or greater toxicity related to prior bevacizumab or daily temozolomide therapy
* Requires therapeutic anti-coagulation with warfarin
* Life expectancy of <12 weeks
* Active malignancy other than basal or squamous cell skin ca or carcinoma in situ of cervix within 5 years
* Subject recruitment and compensation - subjects will be recruited for this study as follows:

  * Upon determination that a subject's tumor histology and/or radiographic findings are compatible with the eligibility criteria of this protocol, the clinical study will be briefly explained to the subject by the subject's physician, who will be a physician at the Brain Tumor Center at Duke.
  * If the subject indicates interest in study participation, subject education sheets and the informed consent document will be provided to the subject as these provide the most comprehensive explanation of the study in lay terms.
  * If the subject shows continued interest, the PI or designee will thoroughly explain the required elements of the consent form and all aspects of the study to the subject including inclusion/exclusion criteria, risks, benefits, and alternatives to study participation.
  * Subjects will not be paid to take part in this research study.

The list of subjects pre-screened will be kept in an Excel spreadsheet in the study coordinator's office. The PC (personal computer) is on the DUHS (Duke University Health System) network protected by a user ID (identifier) and password and the office is locked when it is unoccupied. All screened subjects who are not enrolled in the study will have all identifiers destroyed immediately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peters, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients must have histologically confirmed diagnosis of malignant glioma (Grade 3 or 4 for Phase I and only Grade 4 for Phase II) and radiographic evidence of recurrence or disease progression following prior therapy.
Groups:
- Phase I Dose Escalation: Bevacizumab is to be administered intravenously at 10 mg/kg every other week starting on day 1. Temozolomide is to be administered on a continuous daily dosing schedule at 50 mg/m2/day. Vorinostat (200mg/dose or 400mg/dose) is to be administered daily on days 1-7 and 15-21 of each 28 day cycle. The dose of Vorinostat is escalated in successive 3+3 cohorts of patients to determine the maximum tolerated dose (MTD) of this regimen. The MTD is the dose level at which 0/6 or 1/6 patients experience dose-limiting toxicity (DLT) with at least two patients experiencing DLT at the next higher dose level.
- Phase II: Bevacizumab is to be administered intravenously at 10 mg/kg every other week. Temozolomide is to be administered on a continuous daily dosing schedule at 50 mg/m2/day. Vorinostat is to be administered daily on days 1-7 and 15-21 of each 28 day cycle using the MTD from Phase I.
Period: Overall Study
Arm/Group | Phase I Dose Escalation | Phase II
Started | 9 | 39
Completed | 9 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Escalation | Phase II | Total
Number analyzed (Participants) | 9 | 39 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (14) | 51 (11) | 50 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 15
  Male | 6 | 27 | 33

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Determination of the Maximum Tolerated Dose (MTD)
Description: The MTD is based upon dose-limiting toxicities (DLTs) experienced during Cycle 1 of treatment. The MTD is the dose level at which 0/6 or 1/6 patients experience DLT with at least two patients experiencing DLT at the next higher dose level. Using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, DLTs are defined as: Grade 4 neutropenia lasting greater than 5 days; Grade 3 thrombocytopenia; the occurrence of non-hematologic Grade 3 or greater drug-related adverse events excluding Grade ≥ 3 elevation in alkaline phosphatase, Grade ≥ 3 nausea or vomiting unless occurring despite the use of standard anti-emetics or Grade 3 diarrhea unless occurring despite standard anti-diarrheal therapy; > 14 day delay to re-treat due to failure to resolve drug-related toxicity to re-treatment criteria or pre-treatment baseline.
Time Frame: Cycle 1 (28 days)
Measure: Number; unit: mg
Arm/Group | Phase I Dose Escalation
Number analyzed (Participants) | 9
mg | 400

2. Primary Outcome: Phase II: 6-month Progression-free Survival (PFS)
Description: Phase II: Percentage of participants surviving six months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression according to RANO criteria, or to death due to any cause. Per RANO, progression is a ≥ 25% increase in the sum of the products of perpendicular diameters of enhancing lesions, any new lesion or clinical deterioration.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 39
percentage of participants | 53.8 [37.2 to 67.9]

3. Secondary Outcome: Phase II: Radiographic Response.
Description: The percentage of participants with a complete or partial response as determined by modified Response Assessment in Neuro-Oncology (RANO) criteria. A confirmation of response was not required. Complete Response (CR) was defined as complete disappearance on MR/CT of all enhancing tumor and mass effect, off all corticosteroids (or receiving only adrenal replacement doses) and accompanied by a stable or improving neurologic examination. Partial Response (PR) was defined as greater than or equal to 50% reduction in tumor size on MR/CT by bi-dimensional measurement, on a stable or decreasing dose of corticosteroids and accompanied by a stable or improving neurologic examination. Tumor assessments were done at baseline, the end of the first cycle (4 weeks), then the end of every second cycle (every 8 weeks) thereafter.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 39
percentage of participants | 56 [41 to 71]

4. Secondary Outcome: Phase II: Median Progression-free Survival (PFS)
Description: Phase II: Time in months from the start of study treatment to the date of first progression according to RANO criteria, or to death due to any cause. Per RANO, progression is a ≥ 25% increase in the sum of the products of perpendicular diameters of enhancing lesions, any new lesion or clinical deterioration. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 39
months | 6.7 [4.8 to 9.4]

5. Secondary Outcome: Phase II: Median Overall Survival (OS)
Description: Phase II: Time in months from the start of study treatment to date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 39
months | 12.5 [8.8 to 14.3]

6. Secondary Outcome: Phase II: Number of Patients With Grade 2 or Greater, Treatment-related Toxicities
Description: Phase II: Number of patients with grade 2 or greater, treatment-related toxicities based on Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Phase II
Number analyzed (Participants) | 39
participants | 33

ADVERSE EVENTS:
Time Frame: 3 years
Description: The adverse events for this study were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, and have been converted to CTCAE version 4.0 for entry into ClinicalTrials.gov.
Arm/Group | Phase I Dose Escalation | Phase II
Serious Adverse Events (participants affected / at risk) | 0/9 | 5/39
Other Adverse Events (participants affected / at risk) | 9/9 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalation (N=9) | Phase II (N=39)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Extraocular muscle paresis (Eye disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 3
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalation (N=9) | Phase II (N=39)
Anemia (Blood and lymphatic system disorders) | 6 | 11
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Extraocular muscle paresis (Eye disorders) | 1 | 6
Eye disorders - Other, specify (Eye disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 7 | 19
Diarrhea (Gastrointestinal disorders) | 5 | 24
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 3
Mucositis oral (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 6 | 22
Vomiting (Gastrointestinal disorders) | 4 | 8
Chills (General disorders) | 0 | 2
Edema limbs (General disorders) | 1 | 1
Fatigue (General disorders) | 9 | 32
Fever (General disorders) | 0 | 2
Gait disturbance (General disorders) | 1 | 4
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 2 | 4
Infections and infestations - Other, specify (Infections and infestations) | 0 | 6
Sinusitis (Infections and infestations) | 1 | 4
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 6
Alkaline phosphatase increased (Investigations) | 2 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 9
Blood bilirubin increased (Investigations) | 1 | 7
Creatinine increased (Investigations) | 3 | 8
Neutrophil count decreased (Investigations) | 5 | 17
Platelet count decreased (Investigations) | 8 | 28
White blood cell decreased (Investigations) | 7 | 24
Anorexia (Metabolism and nutrition disorders) | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 23
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 9
Hypernatremia (Metabolism and nutrition disorders) | 2 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 16
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalemia (Metabolism and nutrition disorders) | 3 | 6
Hyponatremia (Metabolism and nutrition disorders) | 1 | 13
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Ataxia (Nervous system disorders) | 1 | 5
Cognitive disturbance (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 2 | 5
Headache (Nervous system disorders) | 7 | 13
Memory impairment (Nervous system disorders) | 1 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 4
Seizure (Nervous system disorders) | 4 | 2
Tremor (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 0 | 2
Confusion (Psychiatric disorders) | 1 | 2
Delayed orgasm (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 2 | 3
Psychosis (Psychiatric disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 5 | 16
Urinary incontinence (Renal and urinary disorders) | 2 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 5 | 8
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes